CLINICAL TRIAL: NCT01608022
Title: A Phase II Trial of PF-00299804 in Patients With Metastatic or Recurrent Squamous Cell Carcinoma of Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0014
Record Dates: First submitted 2012-05-18; First posted 2012-05-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF804 (Experimental)
  Interventions: Drug: PF804

INTERVENTIONS:
Drug: PF804 — 45 mg p.o. daily and continuously (28-day treatment as one treatment cycle)

SUMMARY:
Esophageal cancer (EC) is the eighth most common cause of cancer-related death in the worldwide. Systemic chemotherapy in patients with metastatic EC has limited effectiveness, resulting in a median survival of 8 months to 10months. The low activity and brief duration of benefit for chemotherapy to palliate advanced disease make clear need to identify new active agents.

Epidermal growth factor receptor (EGFR) is often over-expressed, and have been related to poor prognosis in patients with EC. The association between EGFR-activated signaling pathways and tumor cell survival are well documented in many studies. Some EGFR tyrosine kinase inhibitors (TKIs) already showed clinical efficacy against EC. A study with erlotinib showed objective response rate of 15% (2 of 13 patients), but activity was limited to squamous cell type.8 In another study, thirty patients with malignant solid tumor were treated with BIBW2992, irreversible inhibitor of EGFR and HER2, and one of four EC patients achieved partial response.

PF-00299804 is a second-generation quinazoline-based irreversible pan-HER inhibitor. In preclinical studies, PF-00299804 has much lower IC50 values than gefitinib in cell lines engineered to express EGFRvIII mutations (1.2 nM versus 2,700 nM) and produces tumor growth inhibition in gefitinib-resistant xenografts. PF-00299804 reportedly have clinical anti-tumor activity in patients with non-small cell lung cancer and head and neck squamous cell carcinoma with manageable toxicity.

The aim of current trial is to evaluate the antitumor efficacy and safety profile of PF-00299804 and to identify biomarker to predict the tumor response to PF-00299804.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of esophagus
2. Age >= 18
3. ECOG PS 0-2
4. Ineligibility for local therapy (surgery or radiotherapy)
5. Not more than one prior palliative therapy
6. At least one bidimensionally measurable disease as defined by RECIST ver 1.1
7. Adequate organ function for treatment

   * Absolute neutrophil count (ANC)>=1000cells/mm3
   * Platelets >=100000 cells/mm3
   * Estimated creatinine clearance>=50mL/min, or serum creatinine<1.5 x institution upper limit of normal
   * Bilirubin=<1.5 x upper limit of normal(ULN)
   * AST(SGOT)=<2.5 x ULN (5.0xULN if hepatic metastases)
   * ALT(SGPT)=<2.5 x ULN (5.0xULN if hepatic metastases)
   * 12-Lead electrocardiogram(ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
   * QTc interval =<470 msec and without history of Torsades de Points or other symptomatic QTc abnormality
   * LVEF (by MUGA or echocardiogram) of >=50%.
8. The patient has provided signed informed consent and is amenable to compliance with protocol schedules and testing.

Exclusion Criteria:

1. Previous treatment with small molecule EGFR tyrosine kinase inhibitors
2. Two or more previous systemic cytotoxic chemotherapy (Chemotherapy administered with concurrent radiotherapy for local control is not counted)
3. Any major operation or irradiation within 4 weeks of baseline disease assessment
4. Any clinically significant gastrointestinal abnormalities which may impair intake or absorption of the study drug
5. CNS metastasis with continuous corticosteroid use within 4 weeks of baseline disease assessment
6. Patients with known interstitial lung disease
7. Patients with uncontrolled or significant cardiovascular disease (AMI within 12 months,Unstable angina within 6 months, NYHA Class III, IV Congestive heart failure or left ventricular ejection fraction below local institutional lower limit of normal or below 45%, Congenital long QT syndrome, Any significant ventricular arrhythmia, Any uncontrolled second or third degree heart block, Uncontrolled hypertension)
8. Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 5 years prior to study entry.
9. Pregnant or breast-feeding women
10. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation or investigational product administration or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 28th day of every chemotherapy cycle
  Objective Tumor Response will be performed according to the Response Evaluation in Solid Tumor Criteria (RECIST).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea